CLINICAL TRIAL: NCT03306628
Title: Early Carbon Dioxide Laser Therapy for Alleviation of Incisional Scar Burden
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Dr. Hazen is no longer full-time faculty / was not able to find an appropriate PI to take over study.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-01153
Record Dates: First submitted 2017-10-04; First posted 2017-10-11 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Skin Scarring
Keywords: Skin Scarring; keloids; hypertrophic scars; CO2 laser therapy
MeSH Terms: conditions — Cicatrix; Keloid; Cicatrix, Hypertrophic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Laser Therapy (Experimental): a group which will receive laser therapy to one breast incision at the first post-operative visit
  Interventions: Other: CO2 Laser Administration
- Late Laser Therapy (Experimental): a group which will receive laser therapy to one breast incision 6 weeks after surgery
  Interventions: Other: CO2 Laser Administration

INTERVENTIONS:
Other: CO2 Laser Administration — The CO2 fractional laser system will be applied at a pulse energy setting of 50 millijoules and a density of 100 spots/cm2 on one of the breast incisions (either one week after surgery or six weeks after surgery, depending on the randomization group).

SUMMARY:
This is a prospective, randomized pilot study of patients who will undergo either early or late incisional laser therapy after breast reduction surgery to alleviate scar burden at NYU Langone Medical Center. The purpose of this study is to see how well carbon dioxide (CO2) laser therapy works at preventing scar formation after surgery.CO2 laser therapy is currently being used by dermatologists and plastic surgeons to help with scarring after acne and to rejuvenate the face; its benefits are now being explored by medical professionals in dermatology and cosmetic surgery to prevent scarring after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients of all ethnic origins will be considered, although certain ethnic groups will be preferentially excluded more than others such as black and South Asian patients due to our exclusion criteria related to darker skin individuals (see below).
* Patients undergoing bilateral breast reduction surgery

Exclusion Criteria:

* Males will be excluded from this study as male patients rarely undergo breast reduction surgery. When males do undergo breast reduction surgery for gynecomastia, it is often unilateral, and is performed with several techniques and incision types that are not typical employed during female breast reduction. Thus, for this study, only female patients will be considered (see below).
* Any patient enrolled in this study who shows evidence of delayed wound healing, dehiscence, or post operative infection at the first post operative visit will be excluded
* Patients with darker skin (Fitzpatrick IV and above), which is a well-known contraindication to laser therapy
* Pregnant patients
* Patients who have had prior breast surgery
* Patients who have had prior chest/breast irradiation
* Patients with the following diseases which interferes with wound healing: prior hypertrophic scarring/keloids, type I or type II Diabetes Mellitus, autoimmune diseases/collagen vascular diseases
* Patients who are active smokers
* Patients using blood thinners that cannot be stopped
* Patients who have used aspirin within a week of the procedure date

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2019-08-26 (Estimated); Study Completion 2019-08-26 (Estimated)

PRIMARY OUTCOMES:
Change in Vancouver Scar Scale Score | 1 Week to Post Laser 1-Year
  Total of score of each measure below:
  * Pigmentation (0-2) Normal 0 Hypopigmentation 1 Hyperpigmentation 2
  * Vascularity (0-3) Normal 0 Pink 1 Red 2 Purple 3
  * Pliability (0-5) Normal 0 Supple 1 Yielding 2 Firm 3 Banding 4 Contracture 5
  * Height (0-3) Normal (flat) 0 0-2 mm 1 2-5 mm 2 >5 mm 3

CONTACTS AND LOCATIONS:
Overall Officials: Alexes Hazen, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No